CLINICAL TRIAL: NCT01359267
Title: A Pilot Feasibility Study of 99mTc EC DG SPECT/CT Imaging in the Treatment Response Evaluation in Patients With Locally Advanced Head and Neck Cancer
Brief Title: Feasibility of Imaging in the Treatment of Patients With Advanced Head and Neck Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 11-0032
Record Dates: First submitted 2011-05-20; First posted 2011-05-24 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — technetium 99m ethylenedicysteine deoxyglucose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Imaging (Experimental)
  Interventions: Drug: 99mTc-EC-DG

INTERVENTIONS:
Drug: 99mTc-EC-DG — 99mTc-EC-DG will be used before the SPECT/CT scans throughout the study to determine the its effectiveness. 20 mCi of 99mtc-EC-DG will be administered through a vein through a catheter. This will be done before the SPECT/CT scan at 4 weeks and 10 weeks.

SUMMARY:
The purpose of this study is to obtain preliminary information on the potential of 99m Tc-EC-DG SPECT imaging to distinguish cancer from non cancer.

ELIGIBILITY:
Inclusion Criteria:

* Treatment naive patients with histologically proven cancer of the head and neck
* T4 primary tumor (all sites), N2 or N3 locoregional disease (all sites)
* At least one measurable site of disease
* At least 18 years of age
* Karnofsky performance status > or = 70% or ECOG <2
* Able to tolerate SPECT/CT imaging
* Adequate bone marrow function
* Adequate liver function
* Adequate renal function
* Written consent from patients
* Female patients of childbearing potential must have a negative pregnancy test within 0-7 days prior to the first SPECT study

Exclusion Criteria:

* Diabetics with insulin dependence or blood sugar levels >200 mg/dL prior to imaging
* Patient weight above the SPECT/CT table weight limit
* Pregnant and/or lactating female
* Unequivocal demonstration of metastatic disease
* Patients unwilling to or unable to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04-19 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2015-09-15 (Actual)

PRIMARY OUTCOMES:
Persistent Disease within 6 months of CRT | 6 months

SECONDARY OUTCOMES:
Persistent Disease within 2 years of CRT | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States